CLINICAL TRIAL: NCT00261157
Title: Use of Robotic Telerounding After Operative Procedures: Does It Affect Patient Outcomes?
Brief Title: Use of Robotic Telerounding After Operative Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 200412323-1
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2005-12-02 (Estimated); Status verified 2005-11

CONDITIONS: Post-Operative in-Patients
Keywords: nephrectomy; Safety; Laparoscopy; telerounding; prostatectomy

INTERVENTIONS:
Device: InTouch Telerounding Robot

SUMMARY:
This research is being done to test a two-way video system mounted on top of a robot. After surgery the act of seeing and evaluating patients in the hospital is called standard "rounding". This research study will allow doctors to see and speak with their patients using the two-way video system - "telerounding", during their stay at the hospital. The purpose of this study is to assess the safety of telerounding during a patients hospital stay.

Our hypothesis is that post-operative morbidity and the time to identification of post-operative morbidity will not vary with this new method of rounding.

DETAILED DESCRIPTION:
The Department of Urology and the University of California, Davis has made a major commitment to the development of novel applications of advanced telecommunications to the practice of modern health care.

Telemedicine has become an increasingly important although underutilized component of modern healthcare. To date, telemedicine has been limited to physician education in the form of video conferencing for seminars, and to providing specialist consultation in rural medical clinics. However, given the recent technological advances in wireless Internet capabilities and the decreasing cost of these services, we see alternate capabilities for this technology.

As is well known, the act of seeing patients at the bedside while they are hospitalized is called "rounding." For patients that have undergone an elective minimally invasive surgical procedure, such as laparoscopy, hospital stays have become brief events. In fact, the convalescence from these procedures is measured in days rather than weeks. For most individuals, the hospitalization is necessary to allow for the delivery of IV fluids, to check serum chemistries and blood counts while waiting for bowel function to return. To this end, the physician bedside visit is in large part an opportunity to relay information regarding the progress of recovery based on objective laboratory and vital sign measures.

We have developed a video-conferencing system that allows physicians to see and speak with their patients from a remote location (telerounding). In a randomized trial of telerounds versus standard rounds conducted while I was a Urology Fellow at Johns Hopkins, we examined the impact of this form of post-operative management on elements of patient satisfaction with their hospitalization. We found that patients managed with the telerounding system gave higher ratings for their hospitalization than those managed by standard bedside rounds. One such application is the use of teleconferencing as a primary mode of post-operative care management (telerounding). In a prior study we performed at Johns Hopkins, patients expressed higher ratings of satisfaction when the telerounding system was added to usual post-operative care. However, that project was not designed to address the issue of patient safety.

The purpose of the study is to assess if there is a difference in patient outcomes when post-operative patients are managed with "standard rounding" versus "telerounding". Our primary outcome measure is time to recognition of post-operative morbidity. The telerounding system will consist of a wireless Internet-based videoconferencing device mounted on a remotely controlled service robot.

This study will be a prospective, randomized trial. The study population will consist of patients scheduled for laparoscopic radical prostatectomy for the treatment of prostate cancer.

Patients will undergo their scheduled surgery and receive the usual perioperative and immediate post-operative care delivered by the recovery room staff. Once transferred to the patient floor, intervention patients will communicate with their attending physician on a daily basis via the teleconferencing system. Intervention patients will not be seen at the bedside by their attending surgeon. The hospital and resident staff will provide routine daily bedside care. Patients may remove themselves from the study at any time by requesting a bedside visit by the attending physician. The intervention will conclude with either the hospital discharge or identification of a major post-operative morbidity. Intervention arm participants will then participate in a series of focus groups. These sessions will serve as the basis for a detailed qualitative analysis of patient perceptions of this technology and its role in future health care.

ELIGIBILITY:
Inclusion Criteria: Patients, both men and women, undergoing a minimally invasive surgery at the UC Davis Medical Center who are over the age of 18 will be selected. Patients must have an expected hospital stay of greater than 24 hours but less than 72 hours.

Exclusion Criteria: Patients whose anticipated hospital stay exceeds 72 hours will not be included in this study.

-

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2004-04; Study Completion 2005-06

PRIMARY OUTCOMES:
The expected rate of morbidity after a laparoscopic urologic procedure is 16%. Two hundred eighty-four patients are required to detect a 1% difference in morbidity at a 0.05 alpha

CONTACTS AND LOCATIONS:
Overall Officials: Lars Ellison, M.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States